CLINICAL TRIAL: NCT00437541
Title: The Impact of Insulating Domestic Houses on the Health of Occupants: an Intervention Study
Brief Title: Housing, Insulation and Health Study
Acronym: HIHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Insulation study; 01/06/068
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Respiratory Illness; Asthma
Keywords: Insulation; Warmth; Humidity; Damp; Cold; Respiratory; Mould
MeSH Terms: conditions — Asthma; Common Cold

INTERVENTIONS:
Device: Insulation retrofitted into house

SUMMARY:
In six communities we will seek out households where someone who has a history of respiratory problems. For the first winter we will measure temperature and humidity of the house and health of occupants. We will insulate half the houses and the next winter compare them with the uninsulated houses to see if warmer houses improve health.

DETAILED DESCRIPTION:
Damp, cold indoor environments are bad for the health of people who live in them, particularly if they have respiratory problems or are vulnerable, such as the young or the very old. This is a community based study designed to test the hypothesis that insulating domestic houses will make them warmer and that this increase in indoor temperature will improve their health and wellbeing.

Following two pilot studies, the first among older people in city council flats and the second among home owners in Waitara. We have followed the "Waitara model" where community networks will be mobilised to identify households in each community where there is someone with a on going respiratory problem. Seven communities have been selected to help test these hypotheses and have agreed to participate Otara, Gisborne, Mahia/Nuhaka, Taranaki, Porirua, West Coast and Christchurch. Low income areas with high Maori populations have been deliberately selected to maximise the potential health gains.

Two hundred houses in each community will be insulated free of charge to the occupants. The workers who will insulate the homes will be local people employed through the Department of Work and Income (WINZ).

Once the houesholds are selected they will be randomly assigned to intervention or control groups. During the first winter, all 1400 households will be monitored for temperature and humidity and their comfort, health and healthcare utilization will be recorded. Half the households, assigned to the intervention group, will be fully insulated during the spring. The following winter, all the initial measurements taken from both the intervention and control group will be repeated. At the end of the study period, all control houses will be insulated.

This study has developed from a natural intervention being carried out by the Energy Efficiency Conservation Authority (EECA) to insulate domestic houses in New Zealand and is a major collaborative effort, which will shed light on the effectiveness of insulation in improving health and wellbeing. The impact of housing refurbishment on health has not previously been examined. There is considerable government and policy interest in promoting healthy housing and there is strong community interest in ensuring the housing stock is improved in order to lower health risks.

ELIGIBILITY:
Inclusion Criteria:

* Live in Study area
* At least one person in the household must had had respiratory illness within the last year, well members of the same household may also participate
* house currently uninsulated
* interested in taking part in research

Exclusion Criteria:

* Intending to move within study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000
Dates: Start 2001-07; Study Completion 2002-12

PRIMARY OUTCOMES:
Self reported general health, During the first winter post intervention
Indoor temperature and relative humidity, During the first winter post intervention

SECONDARY OUTCOMES:
Energy consumption, During the first winter post intervention
Wheezing, During the first winter post intervention
Days off school and work, During the first winter post intervention
GP visits, During the first winter post intervention
Inpatient hospital admissions, During the first winter post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Philippa L Howden-Chapman, PhD, Study Director — University of Otago; Julian Crane, FRCP, Principal Investigator — University of Otago; Michael G Baker, FRACMA, Principal Investigator — University of Otago; Chris Cunningham, PhD, Principal Investigator — Massey University; Kay Saville-Smith, MA Hons, Principal Investigator — CRESA; Nick Waipara, PhD, Principal Investigator — Landcare Research Limited; Alistair Woodward, PhD, Principal Investigator — University of Otago; Des O'Dea, BSc Hons, Principal Investigator — University of Otago; Tony Blakely, PhD, Principal Investigator — University of Otago; Cheryl Brunton, FAFPHM, Principal Investigator — University of Otago
Locations (8):
- New Zealand (8):
  - Otara Health Inc, Otara, Auckland
  - Crown Public Health, Christchurch, Christchurch
  - Te Iwi O Rakaipaaka, Mahia/Nuhaka, Gisborne
  - Te Wahine O Kahungungu, Mahia/Nuhaka, Gisborne
  - Opotiki Trade Training, Opotiki, Gisborne
  - Te Puni Kokiri, New Plymouth, Taranaki Region
  - Porirua Housing Action Group, Porirua, Wellington Region
  - Maori Womans Welfare League, Rata - Hokitika, West Coast

REFERENCES:
- [Result] Howden-Chapman P, Crane J, Matheson A, Viggers H, Cunningham M, Blakely T, O'Dea D, Cunningham C, Woodward A, Saville-Smith K, Baker M, Waipara N. Retrofitting houses with insulation to reduce health inequalities: aims and methods of a clustered, randomised community-based trial. Soc Sci Med. 2005 Dec;61(12):2600-10. doi: 10.1016/j.socscimed.2005.04.049. Epub 2005 Aug 2. PMID 16061320
- See also: Related Info — http://www.wnmeds.ac.nz/academic/dph/research/housing/index.html